CLINICAL TRIAL: NCT04907331
Title: Comparison of Heterologous Vaccination With an Vaxzevria (ChAdOx1-S) Prime and a Comirnaty (BNT162b2) Boost to Homolog Vaccination
Brief Title: Heterologous SARS-CoV-2 Vaccination With ChAdOx-1 and BNT162b2
Acronym: HeVacc
Status: Unknown | Phase: Phase 2 | Type: Interventional
Last Known Status: Recruiting
Sponsor: Medical University Innsbruck (Other)
Collaborators: Medical University of Graz (Other); Medical University of Vienna (Other)
Responsible Party: Sponsor
Allocation: Randomized | Model: Parallel | Masking: Single | Purpose: Prevention
Other Study IDs: 2021-002171-19
Record Dates: First submitted 2021-05-25; First posted 2021-05-28 (Actual); Last update posted 2021-09-10 (Actual); Status verified 2021-05

CONDITIONS: SARS-CoV2 Infection
MeSH Terms: conditions — COVID-19 | interventions — ChAdOx1 nCoV-19; BNT162 Vaccine

STUDY DESIGN:
Who Masked: Participant
Oversight: Data Monitoring Committee: Yes | FDA-regulated Drug: No | FDA-regulated Device: No | US Export: No

ARMS (3):
- Corminaty twice (Active Comparator): The participants receive Comirnaty twice 3-7 weeks apart
  Interventions: Biological: Comirnaty
- Vaxzevria twice (Active Comparator): The participants receive Vaxzevria twice 12 weeks apart.
  Interventions: Biological: Vaxzevria
- Heterologous (Experimental): The recipients receive Vaxzevria followed by Comirnaty 12 weeks apart
  Interventions: Biological: Vaxzevria; Biological: Comirnaty

INTERVENTIONS:
Biological: Vaxzevria — The participants either receive homologous vaccination with Comirnaty or Vaxzevria as approved or the new heterologous vaccination with Vaxzevria followed by Comirnaty
  Arms: Heterologous; Vaxzevria twice
Biological: Comirnaty — The participants either receive homologous vaccination with Comirnaty or Vaxzevria as approved or the new heterologous vaccination with Vaxzevria
  Arms: Corminaty twice; Heterologous

SUMMARY:
This study will analyze the safety and efficacy of the heterologous vaccination with Vaxzevria followed by Comirnaty. As a control individuals will be vaccinated with Comirnaty or Vaxzevria twice. Each arm will involve 1000 individuals. Endpoints will be the level of antibody and T cell response as well as frequency of vaccine failures.

DETAILED DESCRIPTION:
The immune escape variants are spreading worldwide. Local transmission of the B.1.351 is observed in several European regions while P1 cases are mostly still travel associated. In Austria, there is local transmission of the Czech variant B.1.258 in several regions, while the P1 variant from Brazil plays no role yet. However, B.1.351 local transmission is observed in Tyrol, where 20-30% of SARS-CoV-2 infections were caused by this immune escape variant in January/February 2021, but then controlled but not eliminated by intensive testing. In March and April the largest world-wide outbreak of B.1.1.7 + E484K, also an immune escape variant, was observed in Tyrol. Although, some of the diagnosed cases seemed to be false positive for the E484K mutation, still several hundred have currently already been confirmed, a number that is internationally still unprecedented. It is expected that until the winter infection season, that is likely to hit Europe after a phase of low-level infections in summer, the immune escape variants will make up a substantial portion of SARS-CoV-2 infections in the countries with high seroprevalence after the vaccine campaigns such as Austria. Therefore, the vaccine programs must build up an effective immunity against the wild-type virus as well as the immune escape variants. ChAdOx1-S contributes considerably to the arsenal of vaccines purchased by the European Community. The investigators propose to test whether this vaccine could still be used to build up a cross-protective immunity in the population, when combined with a heterologous boost with the mRNA vaccine BNT162b2. Heterologous prime - boost vaccine regimen including vector vaccines have been broadly used and are generally more effective than homologous vector prime-boost regimen. If ChAdOx1-S followed by BNT162b2 builds up the same or even higher level of cross-neutralizing antibodies as BNT162b2 prime-boost, which is highly likely, the vector vaccine could potentially be included in the program for building a substantial level of cross-immunity against the immune escape variants in the population. Therefore, this study compares the level of cross-neutralizing antibodies induced by classical BNT162b2 and ChAdOx1-S vaccinations with the heterologous prime and boost with ChAdOx1-S followed by BNT162b2, respectively

ELIGIBILITY:
Inclusion Criteria:

1. Subject provides written informed consent
2. Participant is ≥ 18 and ≤ 65 years of age on the day of signing the ICF
3. Individuals that are eligible for vaccination according to the Austrian vaccination plan.
4. Participants that have been vaccinated with either ChAdOx1-S prime within the last 12 weeks or BNT162b2 prime within the last 3 - 6 weeks
5. Subject understands and agrees to comply with study procedures
6. Subject must be willing to be contacted by telephone or willing to complete an eDiary during study participation
7. Female participants of childbearing potential may be enrolled in the study if the participant fulfills all the following criteria:

   * has a negative urine pregnancy test at screening
   * has agreed to practice adequate contraception from providing consent until 3 months after administration of study vaccine
   * is not currently breastfeeding Adequate female contraception is defined as consistent and correct use of an approved contraceptive method, for example:
   * Barrier method (condoms, diaphragm, cervical cap) used in conjunction with spermicide
   * Prescription hormonal contraceptive taken administered via oral (pill), transdermal (patch), subdermal or IM route
   * Intrauterine device
   * Sterilization of a female participant's monogamous male partner prior to study inclusion Cave: periodical abstinence (eg calendar, ovulation, symptothermal,...) and withdrawal are not acceptable methods of contraception.
8. Female participants of non-childbearing potential may be enrolled in the study. Non-childbearing potential is defined as: surgically sterile (history of bilateral dubal ligation, bilateral oophorectomy, hysterectomy) or postmenopausal (amenorrhea for 12 consecutive months prior to Screening without an alternative medical cause).
9. Participants agrees to not donate bone marrow, blood and blood products from the study vaccine administration until 3 months after receiving the study vaccine

Exclusion Criteria:

Participant has already received full vaccination against SARS- CoV-2 2. Prior administration of an investigational coronavirus (SARS- CoV, MERS-CoV) vaccine or current/planned simultaneous participation in another interventional study to either prevent or treat COVID-19 3. Participant has received/plans to receive a non-study vaccine within 14 days prior to or after any dose of IP 4. Participant has a contraindication to IM injections and blood draws (eg, bleeding disorders) 5. Participants has a known or suspected allergy or history of anaphylaxis, urticaria or other significant adverse reactions to vaccines or their excipients (including specifically the excipients of the study vaccine; refer to the IB) 6. Subjects with previous positive PCR-test result for SARS-CoV-2 or positive anti-SARS-CoV-2 N protein antibody test 7. History of leukemia, lymphoma, or underlying bone marrow disorder (eg, myelodysplasia, myeloma, myeloproliferative disorder) or history of bone marrow transplant. 8. Malignancy that required treatment with chemotherapy, immunotherapy, radiation therapy, or other antineoplastic target therapies within 24 months prior to study enrollment. 9. Has participated in an interventional clinical study within 30 days prior to study inclusion

Ages: 18 Years to 65 Years | Sex: All | Healthy Volunteers: Yes
Age Groups: Adult, Older Adult
Enrollment: 3000 (Estimated)
Dates: Start 2021-05-10 (Actual); Primary Completion 2021-11-30 (Estimated); Study Completion 2021-12-30 (Estimated)

PRIMARY OUTCOMES:
Neutralizing antibodies | 10 to 180 days
  in the heterologous arm the levels of neutralizing antibodies are at least as high as in the homologous arms
T cells | 10-180 days
  The level of T cell responses to SARS-CoV-2 S protein epitopes is at leas as high in the heterologous are than in the homologous arms
vaccine failures | 180 days post intervention
  Vaccine failures are not more frequent in the heterologous arm than in the homologous arms.

CONTACTS AND LOCATIONS:
Overall Officials: Dorothee von Laer, MD, Principal Investigator — Medical University Innsbruck
Locations (1):
- Medical University of Innsbruck, Innsbruck, Tyrol, Austria

IPD SHARING:
Plan to Share IPD: No

REFERENCES:
- [Derived] Banki Z, Mateus J, Rossler A, Schafer H, Bante D, Riepler L, Grifoni A, Sette A, Simon V, Falkensammer B, Ulmer H, Neurauter B, Borena W; HEVACC Study Group; Krammer F, von Laer D, Weiskopf D, Kimpel J. Heterologous ChAdOx1/BNT162b2 vaccination induces stronger immune response than homologous ChAdOx1 vaccination: The pragmatic, multi-center, three-arm, partially randomized HEVACC trial. EBioMedicine. 2022 Jun;80:104073. doi: 10.1016/j.ebiom.2022.104073. Epub 2022 May 23. PMID 35617826